CLINICAL TRIAL: NCT05304897
Title: Efficacy and Safety of Platelet-rich Plasma on Bronchopleural Fistula
Brief Title: PRP Efficacy and Safety in BPF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Director of Department of Respiratory Medicine, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20220315
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Bronchopleural Fistula
Keywords: Bronchopleural Fistula; Platelet-rich plasma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRP group (Experimental)
  Interventions: Procedure: PRP treatment

INTERVENTIONS:
Procedure: PRP treatment — PRP treatment for bronchopleural fistula

SUMMARY:
Platelet-rich plasma(PRP), is a concentrate of platelet-rich plasma protein derived from whole blood. The main components of it are platelets, leukocytes and fibrin. Autologous PRP treatment can avoid the immune rejection caused by exogenous growth factor and the spread of disease. Evidence of the efficacy and safety of PRP has been proven in many studies. Bronchopleural fistula (BPF) represents a challenging clinical entity characterized by abnormal communication between the bronchial tree and the pleural space. Respiratory intervention has become one of the most common treatments to fight the disease. Although the short-term occlusion effect of conventional treatment methods of respiratory intervention is relatively easy to achieve, there is great uncertainty in the long-term treatment effect, and long-term large fistulas have little chance of healing. PRP has shown significant efficacy for hyperplastic scar of skin. Correspondingly, PRP will be applied as treatment of BPF to cure fistula.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with aged between 18 to 75
* Subjects diagnosed with bronchopleural fistula (the sizes of the fistulas less than 4mm)
* Subjects willing to accept PRP treatment

Exclusion Criteria:

* Subjects with fistulas larger than 4mm
* Subjects who cannot tolerate bronchoscopy due to severe cardiac disease or other major comorbidities
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-04-16 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Cure rate for bronchopleural fistula | within 4-6 weeks after administration
  Proportion of patients who is no need for endotracheal intervention and with stable clinical symptoms after PRP treatment

SECONDARY OUTCOMES:
the modified Medical Research Council dyspnea scale (mMRC scale) | within 4-6 weeks after administration
  The alleviation or aggravation of dyspnea assessed by the mMRC scale
COPD Assessment Test (CAT) | within 4-6 weeks after administration
  Change of respiratory symptoms and quality of life evaluated by the CAT

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Institute of Respiratory Disease, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No